CLINICAL TRIAL: NCT05328583
Title: A Phase I Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral HRS5685 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral HRS5685 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RetroLead (Shanghai) BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HRS5685-101
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Human Immunodeficiency Virus-1 (HIV-1) Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Treatment group A（Part A） (Experimental): Drug1: HRS5685, dose 1; Drug2: Placebo
  Interventions: Drug: HRS5685；Placebo
- Treatment group B（Part A） (Experimental): Drug1: HRS5685, dose 2; Drug2: Placebo
  Interventions: Drug: HRS5685；Placebo
- Treatment group C（Part A） (Experimental): Drug1: HRS5685, dose 3; Drug2: Placebo
  Interventions: Drug: HRS5685；Placebo
- Treatment group D（Part A） (Experimental): Drug1: HRS5685, dose 4; Drug2: Placebo
  Interventions: Drug: HRS5685；Placebo
- Treatment group E（Part A） (Experimental): Drug1: HRS5685, dose 5; Drug2: Placebo
  Interventions: Drug: HRS5685；Placebo
- Treatment group F（Part A） (Experimental): Drug1: HRS5685, dose 6; Drug2: Placebo
  Interventions: Drug: HRS5685；Placebo
- Treatment group G（Part B） (Experimental): Drug1: HRS5685, dose 3; Drug2: Placebo
  Interventions: Drug: HRS5685；Placebo
- Treatment group H（Part B） (Experimental): Drug1: HRS5685, dose 4; Drug2: Placebo
  Interventions: Drug: HRS5685；Placebo

INTERVENTIONS:
Drug: HRS5685；Placebo — Drug1: HRS5685 Single dose in group A-F and multiple doses in group G-H
  Drug2: Placebo Single dose in group A-F and multiple doses in group G-H

SUMMARY:
This is a randomized, double-blinded, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of single ascending dose (Part A) and multiple ascending dose (Part B) of HRS5685 tablet in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the study protocol;
2. Must be 18 to 45 years of age (inclusive);
3. Body weight of at least 50 kg for male, and 45 kg for female; and Body Mass Index (BMI) within the range of 18 to 28 kg/m2 (inclusive);
4. Physical examination, vital signs, laboratory tests, 12-lead ECG, eGFR (CKD-EPI formula), abdominal ultrasound and chest radiograph are normal or are judged not clinically significant by the investigator;
5. Subjects (including partners) of childbearing potential are willing to useprotocol specified effective methods of contraception from screening to at least 8 months (for female) or 6 months (for male) after the final dose of study drug;

Exclusion Criteria:

1. History or presence of any clinically significant cardiovascular, endocrine, neurological, gastrointestinal, respiratory, hematological, immunological, psychiatric, metabolic disorders or any diseases that may interfere with the study results;
2. Subjects with severe infections, severe trauma or major surgical operation within 3 months before drug administration; or subjects plan to undergo surgery during the trial and within two weeks after the end of trial;
3. Abnormal ECG that is clinically significant, or QTcF< 300 msec or >450 msec for men and >460 msec for women;
4. Positive test result of any of the following at screening: hepatitis B surface antigen (HBsAg), hepatitis C antibody, syphilis, or human immunodeficiency virus (HIV) antibody;
5. Suspected allergy to any ingredient in the study drug;
6. Use of any drug that inhibits or induces hepatic metabolism within 1 month prior to the first dose of study drug;
7. Any condition or disease that affects the absorption, metabolism, and/or excretion of the study drug as judged by the investigator;
8. Use of any prescription or over-the-counter medication, including herbal medications within 1 month prior to the first dose of study drug;
9. Participation in clinical trials of any drug or medical device (except for screening failures) within 3 months before screening, or within 5 half-lives of the drug at screening (whichever is longer);
10. Receiving vaccine(s) within 1 month prior to the first dose of study drug;
11. Donation or loss of blood of ≥ 200 mL within 1 month or of ≥ 400 mL within 3 months prior to the first dose of study drug; or receiving blood transfusion within 8 weeks prior to the first dose of study drug; or have difficulty in venous blood collection, or whose physical condition cannot withstand intensive blood sampling;
12. An average daily smoking of ≥ 5 cigarettes or an average daily alcohol intake of 15 g (15 g alcohol is equivalent to 450 mL beer or 150 mL wine or 50 mL low-alcohol liquor) within 3 months before screening;
13. Subjects who cannot refrain from smoking and alcohol intake from 2 days before the start of study treatment until the last follow-up;
14. Subjects who consume alcoholic beverages, Seville oranges, grapefruit or juices, or products containing caffeine or xanthine (such as coffee, tea, cola drinks and chocolate) from 2 days before the start of study treatment, and those who have special dietary requirements and cannot comply with the unified diet;
15. Subjects with a history of drug abuse, drug dependence, or a positive drugs of abuse test, or a positive alcohol breath test before study drug administration;
16. Pregnant or lactating females;
17. Other conditions judged by the investigator to be not suitable to participate in the trial;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Incidence and severity of adverse events | Up to Day 63 after the last dose

SECONDARY OUTCOMES:
Area under the concentration-time curve during a dosing interval (AUCtau), | Pre-dose up to Day 63 after the last dose
Area under the concentration-time curve from time zero to the last quantifiable time point t (AUC0-t) | Pre-dose up to Day 63 after the last dose
Area under the concentration-time curve extrapolated to infinity (AUC0-inf ) | Pre-dose up to Day 63 after the last dose
Maximum observed concentration (Cmax) | Pre-dose up to Day 63 after the last dose
Time to Maximum observed concentration (Tmax) | Pre-dose up to Day 63 after the last dose
Half-life (t1/2), | Pre-dose up to Day 63 after the last dose
Apparent clearance (CL/F) | Pre-dose up to Day 63 after the last dose
Apparent volume of distribution (Vz/F) | Pre-dose up to Day 63 after the last dose
Trough concentration (Ctrough) | Pre-dose up to Day 63 after the last dose
Accumulation ratio (Rac), | Pre-dose up to Day 63 after the last dose
Renal clearance (CLr) | Pre-dose up to 72 hours post-dose
Cumulative amount of drug excreted (Ae) | Pre-dose up to 72 hours post-dose
Cumulative percentage of dose recovered (fe) | Pre-dose up to 72 hours post-dose

IPD SHARING:
Plan to Share IPD: Undecided